CLINICAL TRIAL: NCT06083194
Title: Non-invasive Evaluation of Muscle Oxidative Capacity. Study of Its Relationship With Muscular Endurance and Fatigue in Patients With Multiple Sclerosis
Brief Title: Evaluation of Muscle Oxidative Capacity Relationship With Muscular Endurance, Fatigue (Multiple Sclerosis).
Acronym: OXYSEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2023 COSTES
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Near infrared spectroscopy (NIRS); Physical capacities; Fatigue; Muscle oxidative capacity; Skeletal muscle mitochondrial capacity; Muscle oxygen consumption; Single-Leg Heel Raise Test; Endurance
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system. It is characterized by different progressive forms with periods of flare-ups interspersed with phases of remission. MS manifests clinically with signs of multiple neurological dysfunctions as well as less specific symptoms such as fatigue, the prevalence of which is found to be high in these patients and is independently associated with an alteration in their quality of life.

Recently, a non-invasive method for assessing maximal muscle oxidative capacity (mVO2) using optical measurement of muscle oxygenation (near-infrared spectroscopy, NIRS) has been described. Measuring tissue light absorption from a skin sensor facing a muscle, makes it possible to distinguish tissue concentrations of oxyhemoglobin (HbO2) and hemoglobin (Hb). The difference in absorbance of Hb and HbO2 corresponds to the balance of O2 supply and consumption in tissue capillaries, allowing calculation of a time constant (kNIRS, min-1) reflecting mitochondrial function.

Current literature provides reference values in young healthy subjects and MS patients. This index could therefore constitute a particularly interesting non-invasive indicator of mitochondrial functioning, usable in the clinic.

DETAILED DESCRIPTION:
Following an arterial occlusion, the rate of decay of the NIRS signal is only dependent on local O2 consumption. Following an exercise increasing the oxygen consumption of the muscle (isometric contractions for 10 to 15 s), carrying out a series of brief occlusions makes it possible to calculate mVO2 (slope of O2 desaturation at each occlusion). mVO2 decreases exponentially with time, allowing calculation of a time constant (kNIRS, min-1) reflecting mitochondrial function. Furthermore, it has been shown that kNIRS correlates with mitochondrial respiration rate measured in oxygraphy (Ryan et al., 2014).

A few studies have focused on the link between maximal muscular oxidative capacity (mVO2), fatigue and muscular endurance in patients with MS. Furthermore, contradictory results have been reported regarding mVO2 in this population, suggesting in one case a higher mVO2 compared to healthy subjects while others observe the opposite. This results in an imprecise assessment of maximum muscle oxidative capacity (mVO2) in MS patients and its relationship with fatigue and muscular endurance in this population. The investigator therefore propose to carry out a prospective interventional study to analyze the relationship between these different parameters. The investigator's hypothesis is the existence of a positive correlation between mVO2 and muscular endurance, and negative with fatigue. This relationship will also be sought 6 months after participants engagement in regular physical activity. Given the accumulation of functional deficits, this approach is focused on preventive medicine, and with the aim of improving the care of these patients.

The statistical analyzes will be carried out with Stata software (version 15; StataCorp, College Station, Texas, USA), considering a risk of two-sided first type error of 5%.

Continuous variables will be presented in the form of mean and standard deviation, according to the normality of their distribution (Shapiro-Wilk test if necessary). In case of non-normality, they will be presented in the form of median, quartiles and extreme values. Qualitative variables will be expressed in numbers and associated percentages.

Graphical representations will, as much as possible, be associated with these analyses.

A description of the deviations from the protocol, the patients distributed according to these deviations and the causes of abandonment will also be carried out. The number of patients included and the inclusion curve will be presented by group.

Patients will be described at inclusion according to the following variables: compliance with eligibility criteria, epidemiological characteristics, clinical characteristics and possible treatments.

The main analysis aiming to investigate the association between maximum muscle oxidative capacity (mVO2) of MS patients assessed by near-infrared spectroscopy (NIRS) and muscular endurance of the gastrocnemius muscles assessed with the unipedal plantar flexion test (Single- Leg standing Heel Raise Test (SLSHR)) will be based on a regression coefficient (Pearson or Spearman with regard to the statistical distribution), interpreted with regard to the recommendations reported in the literature.

The main analysis could be supplemented by a multivariate analysis aimed at taking into account possible confounding factors (including form/type of MS, functional deficits and age); a multiple linear regression will be proposed. The normality of the residuals will be studied; if necessary, a transformation (for example logarithmic) of the dependent variable of the study may be proposed). The results will then be expressed in terms of regression coefficients and 95% confidence interval. A subgroup analysis of the main analysis will be carried out (if possible), according to age, MS, and functional deficits; which will make it possible to evaluate the robustness of the results with regard to the heterogeneity of the sample under study and the possible impact of these variables in addition to the aforementioned multivariate analysis. The maximum muscular oxidative capacity and the muscular endurance of the gastrocnemius muscles could, secondly, be treated and analyzed as categorical data with regard to the work reported in the literature; the study of their relationship will then be analyzed by the most appropriate statistical test. For the study of the relationship between two categorical variables, a chi2 test or a Fisher exact test will be confirmed by presenting the results in terms of absolute difference and 95% confidence interval. The secondary analyzes aiming to study the relationship between the maximum muscular oxidative capacity, the fatigue (FACIT-F questionnaire) and the walking capacity will be based on a regression coefficient (Pearson or Spearman with regard to the statistical distribution) and will be interpreted with regard to the recommendations reported in the literature. The variation in mVO2 at 6 months following the engagement in physical activity [assessed by the variation in energy expenditure (number of METs per week)] will be studied by the paired Student test or the Wilcoxon test; Results will be expressed in terms of effect size and 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Multiple Sclerosis (MS) with a diagnosis established by MRI.
* Patients with a Kurtzke Expanded Disability Status Scale (EDSS) score < 5.
* Body mass index (BMI) < 30 Kg/m².
* Thickness of subcutaneous adipose tissue at the calf ≤ 20 mm.
* MS patients without neurological signs of flare-up since 1 month.
* MS patients who have not had any treatment modification during the last 2 months.
* Subjects affiliated to French health care system (for France).
* Volunteers who have given their written consent.

Exclusion Criteria:

* Patients suffering from progressive psychiatric pathologies (active psychosis, , etc.) or the presence of another serious unstabilized pathology (decompensated heart failure, progressive terminal cancer, etc.).
* People with poorly controlled or unstable cardiovascular disease.
* Major osteoarticular or neurological problems completely preventing the proper performance of the various tests.
* Persons under guardianship, curatorship, deprived of liberty or safeguarding justice.
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis with a Kurtzke Expanded Disability Status Scale (EDSS) score < 5 prospectively assesed for muscle oxidative capacity and muscle endurance.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Maximal muscle oxidative capacity (mVO2) | At the beginning of the protocol inclusion day (to) and at 6 months (t1)
  Maximal muscle oxidative capacity will be measured by near-infrared spectroscopy (NIRS)
Muscular endurance of the gastrocnemius muscles | At the beginning of the protocol inclusion day (to) and at 6 months (t1)
  Muscular endurance of the gastrocnemius muscles, represented by the number of repetitions measured with the Single-Leg Heel Raise Test.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | At the beginning of the protocol inclusion day (to)
  Medical information about the degree of disability patients with Multiple Sclerosis (MS) using the EDSS score; varying between (0 -10). Higher the value higher the disability.
Weight (Kg) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Height (cm) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations.
Waist circumference (cm) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Waist circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Hip circumference (cm) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Hip circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Body Mass Index (Kg/m²) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  BMI will be calculated (weight in kilograms divided by height in meters squared).
Body composition | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Body composition (muscle and fat) will be measured using he Bodystat® Impedance-meter.
Thickness of subcutaneous adipose tissue of the gastrocnemius muscles (mm) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  the measure will be performed using a portable ultrasound machine (Sonobook 6 (CHISON Medical Technologies Co., Ltd.) with a linear probe (40 MHz - 150MHz Linear L7-V). The patient will be in a standing position with the foot placed on a stool so that the thigh is parallel to the ground and the knee joint forms a 90° angle.
Functional capacity | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Functional capacity will be evaluated using the 6-minute walk test.
Gastrocnemius muscle endurance (number of repetitions and time(sec)) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Muscular endurance of the gastrocnemius muscles will be measured with theSingle-Leg Heel Raise Test. Number of repetition will be recorded as well as the time to failure.
Energy expenditure level (MET/minute/week) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Physical activity will be measured using the Global Physical Activity Questionnaire (GPAQ)
Functional Assessment of Chronic Illness Therapy Fatigue Scale | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  The degree of fatigue will be evaluated with the FACIT-F Questionnaire. Score varying between 0 to 52. Higher the score higher the fatigue.
VO2max (maximal oxygen consumption) (mL/Kg/min) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  : VO2max will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum power (Watts) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Maximum power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer
Threshold power (Watts) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Threshold power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer
Maximum heart rate (bpm) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Maximum heart rate will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer
Threshold heart rate (bpm) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Threshold heart will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer
Forced vital Capacity (L and % of the theoretical value) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Forced vital Capacity will be measured with a spirometry test
Forced Expiratory volume (L and % of the theoretical value) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Forced Expiratory volume will be measured with a spirometry test
Tiffeneau ratio (%) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Tiffeneau ratio will be calculated by dividing the Forced Expiratory volume to the Forced vital Capacity.
Ventilatory reserve (%) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  Ventilatory reserve will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Tissue saturation index (kNIRS, min-1) | At the beginning of the protocol inclusion day (to), at 6 months from the inclusion (t1)
  For the determination of mVO2 The patient will be lying down, a cuff (Hokanson SC 12L) will be placed at the level of the thigh, 2 cm from the upper edge of the patella. The NIRS sensor (Portamon, Artinis, Netherlands) will be positioned opposite the body of the two gastrocnemius at the level of its maximum arch, maintained and protected from ambient light by an elastic bandage. The calculation of the absorbances at the 2 wavelengths will be carried out by specific software (Oxysoft) making it possible to display in real time the relative concentrations of Hb and HbO2 and the tissue oxygen saturation (TSI) reflecting muscle O2 saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Fréderic COSTES, Principal Investigator — fcostes@chu-clermontferrand.fr
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Adami A, Rossiter HB. Principles, insights, and potential pitfalls of the noninvasive determination of muscle oxidative capacity by near-infrared spectroscopy. J Appl Physiol (1985). 2018 Jan 1;124(1):245-248. doi: 10.1152/japplphysiol.00445.2017. Epub 2017 Jul 6. No abstract available. PMID 28684592
- [Background] Boushel R, Piantadosi CA. Near-infrared spectroscopy for monitoring muscle oxygenation. Acta Physiol Scand. 2000 Apr;168(4):615-22. doi: 10.1046/j.1365-201x.2000.00713.x. PMID 10759598
- [Background] Edwards T, Pilutti LA. The effect of exercise training in adults with multiple sclerosis with severe mobility disability: A systematic review and future research directions. Mult Scler Relat Disord. 2017 Aug;16:31-39. doi: 10.1016/j.msard.2017.06.003. Epub 2017 Jun 12. PMID 28755682
- [Background] Fromont A, Binquet C, Sauleau EA, Fournel I, Bellisario A, Adnet J, Weill A, Vukusic S, Confavreux C, Debouverie M, Clerc L, Bonithon-Kopp C, Moreau T. Geographic variations of multiple sclerosis in France. Brain. 2010 Jul;133(Pt 7):1889-99. doi: 10.1093/brain/awq134. Epub 2010 Jun 15. PMID 20551111
- [Background] Gelfand JM. Multiple sclerosis: diagnosis, differential diagnosis, and clinical presentation. Handb Clin Neurol. 2014;122:269-90. doi: 10.1016/B978-0-444-52001-2.00011-X. PMID 24507522
- [Background] Hansen D, Feys P, Wens I, Eijnde BO. Is walking capacity in subjects with multiple sclerosis primarily related to muscle oxidative capacity or maximal muscle strength? A pilot study. Mult Scler Int. 2014;2014:759030. doi: 10.1155/2014/759030. Epub 2014 Jan 29. PMID 24624296
- [Background] Harp MA, McCully KK, Moldavskiy M, Backus D. Skeletal muscle mitochondrial capacity in people with multiple sclerosis. Mult Scler J Exp Transl Clin. 2016 Nov 15;2:2055217316678020. doi: 10.1177/2055217316678020. eCollection 2016 Jan-Dec. PMID 28607744
- [Background] Janardhan V, Bakshi R. Quality of life in patients with multiple sclerosis: the impact of fatigue and depression. J Neurol Sci. 2002 Dec 15;205(1):51-8. doi: 10.1016/s0022-510x(02)00312-x. PMID 12409184
- [Background] Kent-Braun JA, Ng AV, Castro M, Weiner MW, Gelinas D, Dudley GA, Miller RG. Strength, skeletal muscle composition, and enzyme activity in multiple sclerosis. J Appl Physiol (1985). 1997 Dec;83(6):1998-2004. doi: 10.1152/jappl.1997.83.6.1998. PMID 9390973
- [Background] Kent-Braun JA, Sharma KR, Miller RG, Weiner MW. Postexercise phosphocreatine resynthesis is slowed in multiple sclerosis. Muscle Nerve. 1994 Aug;17(8):835-41. doi: 10.1002/mus.880170802. PMID 8041390
- [Background] Malagoni AM, Felisatti M, Lamberti N, Basaglia N, Manfredini R, Salvi F, Zamboni P, Manfredini F. Muscle oxygen consumption by NIRS and mobility in multiple sclerosis patients. BMC Neurol. 2013 May 29;13:52. doi: 10.1186/1471-2377-13-52. PMID 23718840
- [Background] Manago MM, Kline PW, Harris-Love MO, Christiansen CL. The Validity of the Single-Leg Heel Raise Test in People With Multiple Sclerosis: A Cross-Sectional Study. Front Neurol. 2021 Jul 21;12:650297. doi: 10.3389/fneur.2021.650297. eCollection 2021. PMID 34354656
- [Background] Motl RW, McAuley E, Sandroff BM, Hubbard EA. Descriptive epidemiology of physical activity rates in multiple sclerosis. Acta Neurol Scand. 2015 Jun;131(6):422-5. doi: 10.1111/ane.12352. Epub 2015 Jan 18. PMID 25598210
- [Background] Nagaraj K, Taly AB, Gupta A, Prasad C, Christopher R. Prevalence of fatigue in patients with multiple sclerosis and its effect on the quality of life. J Neurosci Rural Pract. 2013 Jul;4(3):278-82. doi: 10.4103/0976-3147.118774. PMID 24250159
- [Background] N'Guessan B, Zoll J, Ribera F, Ponsot E, Lampert E, Ventura-Clapier R, Veksler V, Mettauer B. Evaluation of quantitative and qualitative aspects of mitochondrial function in human skeletal and cardiac muscles. Mol Cell Biochem. 2004 Jan-Feb;256-257(1-2):267-80. doi: 10.1023/b:mcbi.0000009874.14649.ca. PMID 14977187
- [Background] Patejdl R, Zettl UK. The pathophysiology of motor fatigue and fatigability in multiple sclerosis. Front Neurol. 2022 Jul 27;13:891415. doi: 10.3389/fneur.2022.891415. eCollection 2022. PMID 35968278
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213
- [Background] Pilutti LA, Sandroff BM, Klaren RE, Learmonth YC, Platta ME, Hubbard EA, Stratton M, Motl RW. Physical Fitness Assessment Across the Disability Spectrum in Persons With Multiple Sclerosis: A Comparison of Testing Modalities. J Neurol Phys Ther. 2015 Oct;39(4):241-9. doi: 10.1097/NPT.0000000000000099. PMID 26247510
- [Background] Razazian N, Kazeminia M, Moayedi H, Daneshkhah A, Shohaimi S, Mohammadi M, Jalali R, Salari N. The impact of physical exercise on the fatigue symptoms in patients with multiple sclerosis: a systematic review and meta-analysis. BMC Neurol. 2020 Mar 13;20(1):93. doi: 10.1186/s12883-020-01654-y. PMID 32169035
- [Background] Rooney S, Wood L, Moffat F, Paul L. Is Fatigue Associated With Aerobic Capacity and Muscle Strength in People With Multiple Sclerosis: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2019 Nov;100(11):2193-2204. doi: 10.1016/j.apmr.2019.06.014. Epub 2019 Aug 6. PMID 31398354
- [Background] Ryan TE, Brizendine JT, McCully KK. A comparison of exercise type and intensity on the noninvasive assessment of skeletal muscle mitochondrial function using near-infrared spectroscopy. J Appl Physiol (1985). 2013 Jan 15;114(2):230-7. doi: 10.1152/japplphysiol.01043.2012. Epub 2012 Nov 15. PMID 23154991
- [Background] Ryan TE, Brophy P, Lin CT, Hickner RC, Neufer PD. Assessment of in vivo skeletal muscle mitochondrial respiratory capacity in humans by near-infrared spectroscopy: a comparison with in situ measurements. J Physiol. 2014 Aug 1;592(15):3231-41. doi: 10.1113/jphysiol.2014.274456. Epub 2014 Jun 20. PMID 24951618
- [Background] Ryan TE, Erickson ML, Brizendine JT, Young HJ, McCully KK. Noninvasive evaluation of skeletal muscle mitochondrial capacity with near-infrared spectroscopy: correcting for blood volume changes. J Appl Physiol (1985). 2012 Jul;113(2):175-83. doi: 10.1152/japplphysiol.00319.2012. Epub 2012 May 10. PMID 22582211
- [Background] Sandroff BM, Klaren RE, Motl RW. Relationships among physical inactivity, deconditioning, and walking impairment in persons with multiple sclerosis. J Neurol Phys Ther. 2015 Apr;39(2):103-10. doi: 10.1097/NPT.0000000000000087. PMID 25742375
- [Background] Sandroff BM, Sosnoff JJ, Motl RW. Physical fitness, walking performance, and gait in multiple sclerosis. J Neurol Sci. 2013 May 15;328(1-2):70-6. doi: 10.1016/j.jns.2013.02.021. Epub 2013 Mar 21. PMID 23522499
- [Background] Sumner MD, Beard S, Pryor EK, Das I, McCully KK. Near Infrared Spectroscopy Measurements of Mitochondrial Capacity Using Partial Recovery Curves. Front Physiol. 2020 Feb 14;11:111. doi: 10.3389/fphys.2020.00111. eCollection 2020. PMID 32116804
- [Background] Trapp BD, Peterson J, Ransohoff RM, Rudick R, Mork S, Bo L. Axonal transection in the lesions of multiple sclerosis. N Engl J Med. 1998 Jan 29;338(5):278-85. doi: 10.1056/NEJM199801293380502. PMID 9445407
- [Background] Zoll J, Bouitbir J, Sirvent P, Klein A, Charton A, Jimenez L, Peronnet FR, Geny B, Richard R. Apparent Km of mitochondria for oxygen computed from Vmax measured in permeabilized muscle fibers is lower in water enriched in oxygen by electrolysis than injection. Drug Des Devel Ther. 2015 Jul 13;9:3589-97. doi: 10.2147/DDDT.S81891. eCollection 2015. PMID 26203225